CLINICAL TRIAL: NCT06689722
Title: Investigation of the Effectiveness of Chiropractic Treatment Applied Together With Ergonomics Education in Factory Workers With Nonspecific Neck Pain: A Randomized Study
Brief Title: Effectiveness of Chiropractic Treatment Applied Together With Ergonomics Education in Factory Workers With Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uskudar University (Other)
Responsible Party: Principal Investigator, Dr. Öğr. Üyesi Ömer Şevgin, Asst. Prof. Dr., Uskudar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Uskudar14
Record Dates: First submitted 2024-11-12; First posted 2024-11-14 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Neck Pain; Work-related Illness
Keywords: chiropractic; occupational diseases
MeSH Terms: conditions — Neck Pain; Occupational Diseases | interventions — Manipulation, Chiropractic; salicylhydroxamic acid; Ergonomics

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- chiropractic (Experimental): chiropractic practices
  Interventions: Other: chiropractic; Other: ergonomics
- placebo (Sham Comparator): sham manipulation applications
  Interventions: Other: sham; Other: ergonomics
- control (Active Comparator): those who did not receive any intervention
  Interventions: Other: ergonomics

INTERVENTIONS:
Other: chiropractic — Chiropractic practice was applied using the diversified technique, which is one of the types of chiropractic techniques.
  Arms: chiropractic
Other: sham — The patient was asked if he/she had any pain or other complaints during the trial mobilization. High-velocity, low-amplitude impulses were applied to the inferior and lateral directions for patients who did not describe any complaints.
  Arms: placebo
Other: ergonomics — Ergonomics training will be given to each of the control group participants individually. The content of this training will include "what is ergonomics, the purpose of ergonomics, musculoskeletal diseases in employees, work-related musculoskeletal risk fa

SUMMARY:
The aim of this study is to investigate the effectiveness of chiropractic treatment combined with ergonomic training in factory workers with nonspecific neck pain.

DETAILED DESCRIPTION:
The study was planned as a randomized controlled study. Workers between the ages of 18-60 who are working in a heat treatment factory in izmir and experiencing non-specific neck pain will be included in the study. The factory workers included in the study will be divided into three by simple random method. The groups will be called chiropractic, placebo and control groups. All participants will be given ergonomic training before the treatment. The chiropractic group will be applied 2 days a week. The placebo group will also be applied sham manipulation 2 days a week. No intervention will be made in the control group. In order to collect data from the participants; Visual Analog Scale, Neck Disability Questionnaire and Bournemouth will be used for pain and pain-related dysfunctions, and Pittsburgh Sleep Quality Questionnaire will be used to determine sleep quality. These questionnaires will be repeated before starting the study and at the end of the study.

ELIGIBILITY:
Inclusion criteria:

* Being between 18-65 years of age,
* Having neck pain for the last 3 months,
* Neck pain being 4 or higher on the Visual Analog Scale

Exclusion criteria:

* Having undergone surgery in the last 6 months,
* Not being cooperative,
* Presence of psychological problems,
* Neck pain being of radicular or neurological origin,
* Presence of a systemic or metabolic disease such as cancer, Instability in the neck,
* Vertebro-basilar insufficiency

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2024-11-15 (Actual); Primary Completion 2024-12-25 (Actual); Study Completion 2025-01-02 (Actual)

PRIMARY OUTCOMES:
The Pittsburgh Sleep Quality Index (PSQI) | 5 weeks
  Pittsburgh Sleep Quality Index; It evaluates sleep duration, sleep disturbance, sleep efficiency, subjective sleep quality, sleep medication use, daytime dysfunction, and sleep delay and consists of a total of 24 questions. 19 of them are self-report scales and 5 of them consist of questions to be answered by a friend or spouse. There are 7 components with 18 questions scored in the scale, and each component is evaluated between 0 and 3 points. The total score ranges from 0 to 21, and 5 or more is an indicator of "poor sleep quality".
Neck Pain Disability Index Questionnaire | 5 weeks
  The scale includes 10 titles. It includes pain sensitivity, heavy lifting, personal hygiene, reading, sleep, headache, concentration, work, driving, social activities. There are 6 answer options according to the severity of the limitation or pain. Scoring is between 0 and 5. The highest score is 50 and the least is 0. The neck disability level classification according to the total score is as follows 0-4: no restrictions 5-14: mild limitation 15-24: moderate limitation 25-34: severe limitation 34 and up: completely restricted
Bournemouth Neck Pain Survey | 5 weeks
  The survey consists of 7 questions. In addition to questions about pain and disability, it also includes questions about psychosocial issues. Each question is scored between 0 and 10. The highest score is 70, with a higher score indicating a higher level of disability. The content of the survey consists of variables that must be questioned for individuals with neck pain, such as pain severity, the effect of pain on daily life activities and social life, anxiety-depression level, kinesiophobia and coping with pain.

CONTACTS AND LOCATIONS:
Overall Officials: Deniz Balıkçı, Study Chair — Bahçeşehir University
Locations (1):
- Kemalpaşa Heat treatment factory, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pehlevan E, Sevgin O. Effect of exercise given to factory workers with ergonomics training on pain and functionality: A randomized controlled trial. Work. 2024;78(1):195-205. doi: 10.3233/WOR-230663. PMID 38701125
- [Background] Zengi H, Safran EE, Sevgin O. The effect of home exercises with kinesiotaping on pain, functionality, and work performance in bus drivers with non-specific neck pain. J Back Musculoskelet Rehabil. 2024;37(6):1617-1630. doi: 10.3233/BMR-240001. PMID 38943382
- [Background] Chaibi A, Allen-Unhammer A, Kopke Vollestad N, Russell MB. Chiropractic spinal manipulative therapy for acute neck pain: A 4-arm clinical placebo randomized controlled trial. A prospective study protocol. PLoS One. 2023 Dec 7;18(12):e0295115. doi: 10.1371/journal.pone.0295115. eCollection 2023. PMID 38060549